CLINICAL TRIAL: NCT03591354
Title: An Extension Study of t:Slim X2 With Control-IQ Technology
Brief Title: The International Diabetes Closed Loop (iDCL) Trial: Clinical Acceptance of the Artificial Pancreas (DCLP3 Extension)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other); Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCLP3 Extension; UC4DK108483 (NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-07-19 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Type 1 Diabetes Mellitus; Insulin Pump; Continuous Glucose Monitor (CGM); Closed Loop Control (CLC); Sensor-Augmented Pump (SAP)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of 3 months at home closed loop system vs. predictive-low glucose suspend.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Closed Loop Control (CLC) (Experimental): Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 Continuous Glucose Monitor (CGM) for 3 months.
  Objective 1: This arm is participants who had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial)
  Objective 2: This arm is participants who had 6 months of sensor-augmented pump (SAP) in the primary trial (DCLP3 Pivotal Trial)
  Objective 3: This arm is participants who had 3 months of CLC in the extension trial (DCLP3 Extension) will continue use of the Control-IQ Technology & Dexcom G6 CGM until the product is commercially available.
  Interventions: Device: t:slim X2 with Control-IQ Technology & Dexcom G6 CGM
- Predictive-Low Glucose Suspend (PLGS) (Active Comparator): Participants randomized to Predictive-Low Glucose Suspend (PLGS) will use the t:slim X2 with Basal-IQ & Dexcom G6 CGM for 3 months.
  Objective 1: This arm is participants who had 6 months of PLGS in the primary trial (DCLP3 Pivotal Trial)
  Objective 2: This arm is not applicable to objective 2
  Objective 3: This arm is participants who had 3 months of PLGS in the extension trial (DCLP3 Extension) will continue use of the Control-IQ Technology & Dexcom G6 CGM until the product is commercially available.
  Interventions: Device: t:slim X2 with Basal-IQ & Dexcom G6 CGM

INTERVENTIONS:
Device: t:slim X2 with Control-IQ Technology & Dexcom G6 CGM — Participants will use the Tandem t:slim X2 insulin pump with Control-IQ Technology & Dexcom G6 CGM for 3 months.
  Arms: Closed Loop Control (CLC)
Device: t:slim X2 with Basal-IQ & Dexcom G6 CGM — Participants will use a Tandem t:slim X2 insulin pump with Basal-IQ and a study CGM (Dexcom G6) for 3 months.
  Arms: Predictive-Low Glucose Suspend (PLGS)

SUMMARY:
This is a 3-month extension study (DCLP3 Extension) following a primary trial (DCLP3 or NCT03563313) to assess efficacy and safety of a closed loop system (t:slim X2 with Control-IQ Technology) in a large randomized controlled trial. Upon completion of the NIH 3-month extension study, subjects will be invited to participate in a continued use phase with Control-IQ Technology, funded by Tandem Diabetes Care, until the equipment has received FDA approval for commercial use.

DETAILED DESCRIPTION:
Participants in the 6 month primary trial (DCLP3) will be invited to continue in this 3-month extension study (DCLP3 Extension) following completion of the primary trial. The closed-loop control (CLC) Intervention Group participants from the primary trial will be randomly assigned to continue CLC or to switch to Predictive Low-Glucose Suspend (PLGS) therapy with t:slim X2 with Basal-IQ and Dexcom G6 for 3 months. The Sensor-Augmented Pump (SAP) Control Group participants from the primary trial will be assigned to CLC using t:slim X2 with Control-IQ Technology and Dexcom G6 (CGM) for 3 months. Upon completion of the extension study, subjects will be invited to participate in continued use of the Control-IQ Technology until the equipment has received FDA approval for commercial use.

This extension phase has two separate objectives:

Objective 1: Among participants who used CLC in the primary trial: the primary efficacy outcome for the randomized controlled trial (RCT) is time in target range 70-180 mg/dL measured by CGM in CLC group vs. PLGS group over 3 months. Safety outcomes also will be assessed Objective 2: Among participants who used SAP in the primary trial: the primary outcome is to obtain additional safety data. Efficacy also will be assessed as a pre-post within participant analysis

Note: Primary Trial (DCLP3) is NCT03563313

ELIGIBILITY:
Inclusion Criteria:

1. Successful completion of the original 6-month RCT within the prior 14 days
2. For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
3. For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact the participant in case of an emergency.
4. Willingness to not use a personal CGM for the duration of the study
5. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol
6. Willingness to use only lispro (Humalog) or aspart (Novolog), and to use no other insulin during the study.
7. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial

Exclusion Criteria

1. Concurrent use of any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
2. Hemophilia or any other bleeding disorder
3. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
4. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
5. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., Dexcom, Inc., or TypeZero Technologies, LLC, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia
Locations (7):
- United States (7):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - Harvard University (Joslin Diabetes Center), Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Time Frame: Generally, data will be made available after the primary publications of each study.
Access Criteria: The Data Sharing Agreements will be formulated by the Steering Committee in collaboration with the NIH Project Scientist Program Official.
  In addition, under special arrangements, complete data sets will be provided to industry partners who would use the data for regulatory clearance (PMA - pre-market approval) of the tested artificial pancreas system. This will be done in response to the specific requirements of RFA-DK-14-024 for this project to "...generate data able to satisfy safety and efficacy requirements by regulatory agencies regarding the clinical testing of artificial pancreas device systems in the target population of people with type 1 diabetes."

REFERENCES:
- [Derived] Levy CJ, O'Malley G, Raghinaru D, Kudva YC, Laffel LM, Pinsker JE, Lum JW, Brown SA; iDCL Trial Research Group. Insulin Delivery and Glucose Variability Throughout the Menstrual Cycle on Closed Loop Control for Women with Type 1 Diabetes. Diabetes Technol Ther. 2022 May;24(5):357-361. doi: 10.1089/dia.2021.0431. Epub 2022 Feb 21. PMID 35099294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Objective 1 (Primary): Participants with 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial) were randomized to either CLC or PLGS with outcomes evaluated during the 3 mo extension.
  Objective 2: Participants with 6 mos of SAP in the primary trial (DCLP3 Pivotal Trial) were then transitioned to CLC during the 3-mo extension.
  Objective 3: All participants who completed the initial 3 mos of the extension trial continued use of CLC until the system was commercially available.
Groups:
- Closed Loop Control (CLC): Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 3 months. Participants in this arm had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm are analyzed as part of the Objective 1 of the trial to compare CLC vs PLGS for 3 months following the use of 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial).
  Participants in this arm will continue to use CLC through commercial availability of the device after completion of the 3 months extension (Objective 3 of the trial).
- Predictive-Low Glucose Suspend (PLGS): Participants randomized to Predictive-Low Glucose Suspend (PLGS) arm will use the t:slim X2 with Basal-IQ & Dexcom G6 CGM for 3 months. Participants in this arm had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm are analyzed as part of the Objective 1 of the trial to compare CLC vs PLGS for 3 months following the use of 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial).
  Participants in this arm will use CLC through commercial availability of the device after completion of the 3 months extension (Objective 3 of the trial).
- SAP to CLC Group: Participants in this arm were transitioned to CLC (t:slim X2 with Control-IQ Technology & Dexcom G6 CGM) after the extension began. Participants in this arm had previously been randomized to Sensor-Augmented Pump (SAP) in the primary trial (DCLP3 Pivotal Trial). This arm met Objective 2 of the study and was not compared to the CLC and PLGS groups that were randomized during the extension.
  Participants in this arm will continue to use CLC through commercial availability of the device after the completion of the 3 months extension (Objective 3 of the trial).
Period: Overall Study
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Started | 54 | 55 | 55
Completed | 54 | 55 | 55
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Predictive-Low Glucose Suspend (PLGS): Participants randomized to Predictive-Low Glucose Suspend (PLGS) arm will use the t:slim X2 with Basal-IQ & Dexcom G6 CGM for 3 months. Participants in this arm had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm are analyzed as part of the Objective 1 of the trial to compare CLC vs PLGS for 3 months following the use of 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial).
  Participants in this arm will use CLC through commercial availability of the device after the 3 months extension (Objective 3 of the trial).
- SAP to CLC Group: Participants in this arm were transitioned to CLC (t:slim X2 with Control-IQ Technology & Dexcom G6 CGM) after the extension began. Participants in this arm had previously been randomized to Sensor-Augmented Pump (SAP) in the prior Pivotal Trial. This arm was not compared to the randomized groups CLC and PLGS that were randomized during the extension. This group met Objective 2 of the study.Participants in this arm will continue to use CLC through commercial availability of the device after the 3 months extension
- Total: Total of all reporting groups
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group | Total
Number analyzed (Participants) | 54 | 55 | 55 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (14) | 34 (17) | 34 (17) | 33 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 30 | 83
  Male | 26 | 30 | 25 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 46 | 46 | 52 | 144
  Race: Non-White | 7 | 7 | 3 | 17
  Race: Did Not Answer | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 54 | 55 | 55 | 164
Diabetes duration [Median (Inter-Quartile Range); unit: years] | 18 [8 to 29] | 16 [7 to 31] | 16 [6 to 23] | 17 [8 to 29]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26 [23 to 30] | 25 [23 to 29] | 26 [22 to 29] | 25 [23 to 29]
Annual household income [Count of Participants; unit: Participants]
  <$50,000 | 5 | 5 | 2 | 12
  $50,000 to < $100,000 | 8 | 13 | 18 | 39
  >= $100,000 | 29 | 26 | 30 | 85
  Did Not Answer | 12 | 11 | 5 | 28
Highest education level [Count of Participants; unit: Participants]
  Less than a bachelor's degree | 8 | 8 | 12 | 28
  Bachelor's degree | 26 | 23 | 21 | 70
  Advanced degree | 19 | 24 | 22 | 65
  Did Not Answer | 1 | 0 | 0 | 1
Insurance [Count of Participants; unit: Participants]
  Private Insurance | 49 | 51 | 50 | 150
  Other Insurance | 2 | 3 | 4 | 9
  No Insurance | 2 | 0 | 0 | 2
  Did Not Answer | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time in Target Range
Description: The primary exploratory outcome is time in target range 70-180 mg/dL measured by CGM comparing the randomized groups CLC vs PLGS. Results from SAP to CLC group is also included here without the primary intention of comparing to CLC vs PLGS groups.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time in range | 67.6 (12.6) | 60.4 (17.1) | 69 (11)
Statistical Analysis 1: Comparison: Closed Loop Control (CLC) vs Predictive-Low Glucose Suspend (PLGS); Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: CGM Time Above 180
Description: CGM-measured % above 180 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 31 (13) | 38 (18) | 29 (11)

3. Secondary Outcome: CGM Mean Glucose
Description: CGM-measured mean glucose
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
mg/dL | 160 (20) | 170 (30) | 158 (17)

4. Secondary Outcome: CGM Time Below 70
Description: CGM-measured % below 70 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 0.53 (0.34) | 0.59 (0.37) | 1.76 (1.07)

5. Secondary Outcome: CGM Time Below 54
Description: CGM-measured % below 54 mg/dL
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 0.2 [0.07 to 0.48] | 0.22 [0.06 to 0.46] | 0.19 [0.08 to 0.36]

6. Secondary Outcome: CGM Time in Range 70-140 mg/dL
Description: CGM-measured % in range 70-140 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 42 (12.5) | 37.1 (14.2) | 45 (10)

7. Secondary Outcome: Coefficient of Variation
Description: CGM measured glucose variability measured with the coefficient of variation (CV)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage SD of Mean
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage SD of Mean | 34 (4) | 35 (5) | 35 (5)

8. Secondary Outcome: Standard Deviation
Description: CGM measured glucose variability measured with the standard deviation (SD)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
mg/dL | 55 (12) | 60 (15) | 56 (12)

9. Secondary Outcome: CGM Time Below 60
Description: CGM-measured % below 60 mg/dL
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 0.43 [0.19 to 0.97] | 0.46 [0.17 to 0.96] | 0.51 [0.30 to 0.78]

10. Secondary Outcome: LBGI
Description: Low blood glucose index by CGM with higher index indicating higher risk of hypoglycemia. Values <1 suggest minimal risk. Index of risk of low blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Gonder-Frederick LA, Young-Hyman D, Schlundt D, Clarke WL: Assessment of risk for severe hypoglycemia among adults with IDDM: validation of the low blood glucose index. Diabetes Care 21:1870-1875, 1998)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
index | 0.53 (0.34) | 0.59 (0.37) | 0.54 (0.24)

11. Secondary Outcome: CGM Hypoglycemia Events
Description: CGM-measured events of at least 15 consecutive minutes <70 mg/dL
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Events per Week
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events per Week | 3.0 [1.5 to 4.9] | 3.1 [1.6 to 5.3] | 3.8 [2.5 to 4.8]

12. Secondary Outcome: CGM Time >250
Description: CGM-measured % >250 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 7 (6.5) | 13.6 (12.4) | 7.8 (6.6)

13. Secondary Outcome: CGM Time >300
Description: CGM-measured % >300 mg/dL
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- SAP to CLC: Participants in this arm were transitioned to CLC (t:slim X2 with Control-IQ Technology & Dexcom G6 CGM) after the extension began. Participants in this arm had previously been randomized to Sensor-Augmented Pump (SAP) in the primary trial (DCLP3 Pivotal Trial). This arm met Objective 2 of the study and was not compared to the CLC and PLGS groups that were randomized during the extension.
  Participants in this arm will continue to use CLC through commercial availability of the device after the completion of the 3 months extension (Objective 3 of the trial).
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC
Number analyzed (Participants) | 54 | 55 | 55
percentage of time | 2.3 (3.4) | 5.2 (6.3) | 2.7 (3.5)

14. Secondary Outcome: HBGI
Description: High blood glucose index by CGM with higher values indicating higher risk of hyperglycemia. Index of risk of high blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Kumar A, Gonder-Frederick L, Clarke WL. Algorithmic evaluation of metabolic control and risk of severe hypoglycemia in type 1 and type 2 diabetes using self-monitoring blood glucose data. Diabetes Technol Ther 2003;5:817-828pmid:14633347)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
index | 6.4 (3.1) | 9.2 (5.3) | 6.6 (3.0)

15. Secondary Outcome: HbA1c at 13 Weeks
Description: HbA1c at 13 weeks.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: % of glycated hemoglobin
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
% of glycated hemoglobin | 7.18 (0.80) | 7.53 (1.14) | 7.09 (0.74)

16. Secondary Outcome: HbA1c <7.0% at 13 Weeks
Description: HbA1c <7.0% at 13 weeks.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 23 | 15 | 26

17. Secondary Outcome: HbA1c <7.5% at 13 Weeks
Description: HbA1c <7.5% at 13 weeks.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Groups:
- SAP-CLC Group: Participants in this arm were transitioned to CLC (t:slim X2 with Control-IQ Technology & Dexcom G6 CGM) after the extension began. Participants in this arm had previously been randomized to Sensor-Augmented Pump (SAP) in the primary trial (DCLP3 Pivotal Trial). This arm met Objective 2 of the study and was not compared to the CLC and PLGS groups that were randomized during the extension.
  Participants in this arm will continue to use CLC through commercial availability of the device after the completion of the 3 months extension (Objective 3 of the trial).
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP-CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 35 | 32 | 39

18. Secondary Outcome: HbA1c Change From Baseline to 13 Weeks >0.5%
Description: HbA1c change from baseline to 13 weeks >0.5%.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 1 | 2 | 14

19. Secondary Outcome: HbA1c Change From Baseline to 13 Weeks >1.0%
Description: HbA1c change from baseline to 13 weeks >1.0%.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 0 | 0 | 5

20. Secondary Outcome: HbA1c Relative Change From Baseline to 13 Weeks >10%
Description: HbA1c relative change from baseline to 13 weeks >10%.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 0 | 0 | 8

21. Secondary Outcome: HbA1c Change From Baseline to 13 Weeks >1.0% or HbA1C <7.0% at 13 Weeks
Description: HbA1c change from baseline to 13 weeks >1.0% or HbA1c <7.0% at 13 weeks.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 23 | 15 | 30

22. Secondary Outcome: HFS-II Adult
Description: Fear of Hypoglycemia Survey (HFS-II) total score and 3 sub scales (5 point scale with never to almost always)
  For adults, teens and parents items on this survey are rated on a 5 point Likert scale from never (0) to almost always (4). The survey is scored by summing item responses. Fear of Hypoglycemia Survey (HFS-II) for adults has a total score that is summed from the two subscale scores (33 items) and ranges from 0 to 132 with higher scores indicating greater degrees of fear of hypoglycemia.
Time Frame: 13 weeks
Population: Adults
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC
Number analyzed (Participants) | 40 | 42 | 41
total score on a scale | 29 (11) | 35 (16) | 33 (14)

23. Secondary Outcome: HFS-II Teen
Description: Fear of Hypoglycemia Survey (HFS-II) total score and 3 sub scales (5 point scale with never to almost always)
  For adults, teens and parents items on this survey are rated on a 5 point Likert scale from never (0) to almost always (4). The survey is scored by summing item responses.The teen survey has a total of 25 items and the range of Total scores is 0 to 100.
Time Frame: 13 weeks
Population: Teens
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 14 | 13 | 12
total score on a scale | 35 (9) | 30 (12) | 30 (13)

24. Secondary Outcome: HFS-II Parents
Description: Fear of Hypoglycemia Survey (HFS-II) total score and 3 sub scales (5 point scale with never to almost always)
  For adults, teens and parents items on this survey are rated on a 5 point Likert scale from never (0) to almost always (4). The parent version of the survey has a total of 26 items with Total scores that range from 0 to 108.
Time Frame: 13 weeks
Population: Parent
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 14 | 13 | 12
total score on a scale | 35 (12) | 40 (18) | 37 (14)

25. Secondary Outcome: Hyperglycemia Avoidance Scale
Description: Hyperglycemia Avoidance Scale total score is the sum of 21 items rated on a 4 point Likert scale from 0 (never) to 4 (almost always) and ranges from 0 to 84 with a higher score indicating greater degrees of avoiding hyperglycemia.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 53
total score on a scale | 37 (9) | 37 (11) | 36 (10)

26. Secondary Outcome: Diabetes Distress Scale
Description: Diabetes Distress Scale for adults has 28 items rated on a 6 point Likert scale that ranges from 1 (not a problem) to 6 (a very serious problem). The total score is the mean of the sum of responses and ranges from 1 to 6 where a higher score indicates greater degrees of diabetes distress.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP-CLC Group
Number analyzed (Participants) | 54 | 55 | 53
total score on a scale | 1.8 (0.7) | 1.7 (0.7) | 1.7 (0.7)

27. Secondary Outcome: Hypoglycemia Confidence Scale
Description: Hypoglycemia Confidence Scale has 9 items which are self-rated on a 4-point Likert Scale ranging from 1 (not confident at all) to 4 (very confident) with higher scores indicating higher confidence in dealing with hypoglycemia. A single score is computed by calculating the mean of the sum of all items and ranges from 1 to 4.
Time Frame: 13 weeks
Population: Reporting first item on the scale: exercise
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Closed Loop Control (CLC): Participants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 3 months. Participants in this arm had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm are analyzed as part of the Objective 1 of the trial to compare CLC vs PLGS for 3 months following the use of 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm will continue to use CLC through commercial availability of the device after the 3 months extension (Objective 3 of the trial).
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 53
score on a scale | 2.0 [1 to 4] | 2.1 [2 to 4] | 1.9 [1 to 4]

28. Secondary Outcome: Clarke Hypoglycemia Awareness Scores
Description: Clarke Hypoglycemia Awareness Scores (0-7 score with higher scores associated with impaired awareness)
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 53
total score on a scale | 1 [0 to 3] | 1 [1 to 3] | 1 [0 to 3]

29. Secondary Outcome: INSPIRE Survey Scores- Adults
Description: The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems: Perceptions, Ideas, Reflections, Expectations (INSPIRE). Survey total scores are computed by calculating the mean of the sum of all item ratings then multiplying the mean by 25 to scale the score to a range from 0 to 100. Higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The Adult survey has 22 items.
Time Frame: 13 weeks
Population: Adults
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 40 | 42 | 41
total score on a scale | 87 (13) | 87 (13) | 84 (17)

30. Secondary Outcome: INSPIRE Survey Scores- Teens
Description: The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems: Perceptions, Ideas, Reflections, Expectations (INSPIRE). Survey total scores are computed by calculating the mean of the sum of all item ratings then multiplying the mean by 25 to scale the score to a range from 0 to 100. Higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The Teens/Adolescents survey has 17 items.
Time Frame: 13 weeks
Population: Teens
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 14 | 13 | 12
total score on a scale | 80 (16) | 89 (15) | 77 (16)

31. Secondary Outcome: INSPIRE Survey Scores- Parents
Description: The INSPIRE questionnaire assesses user expectations and experiences with Insulin Delivery Systems: Perceptions, Ideas, Reflections, Expectations (INSPIRE). Survey total scores are computed by calculating the mean of the sum of all item ratings then multiplying the mean by 25 to scale the score to a range from 0 to 100. Higher scores indicate a more positive perception of insulin delivery systems. Items are rated on a 5 point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). The Parent survey has 21 items.
Time Frame: 13 weeks
Population: Parent.
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 14 | 13 | 12
total score on a scale | 86 (17) | 87 (13) | 86 (11)

32. Secondary Outcome: System Usability Scores (SUS)
Description: System Usability Scores (SUS)-composite score from 0 to 100 with higher scores indicating better perceived usability
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 54 | 53
total score on a scale | 85 (12.3) | 86.6 (11.3) | 85.2 (16.9)

33. Secondary Outcome: Technology Acceptance Questionnaire
Description: Technology Acceptance Survey measures the user's perceptions regarding the burdens and the barriers associated with a technology with a higher score indicates increased technology acceptance. There total score uses 37 items with items are rated on a 5 point scale ranging from 1 (strongly disagree) to 5 (strongly agree) for total score range of 37-185.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 54 | 53
total score on a scale | 151 (17) | 149 (25) | 145 (28)

34. Secondary Outcome: Total Daily Insulin
Description: Total Daily Insulin (units/kg)
Time Frame: 13 weeks
Population: Data not available in all participants
Measure: Median (Inter-Quartile Range); unit: Units of insulin per kg
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 53
Units of insulin per kg
  Baseline | 0.59 [0.49 to 0.86] | 0.68 [0.46 to 0.93] | 0.62 [0.52 to 0.9]
  At 13-week Follow Up: number analyzed (Participants) | 54 | 55 | 52
  At 13-week Follow Up | 0.62 [0.50 to 0.84] | 0.67 [0.48 to 0.88] | 0.64 [0.52 to 0.86]

35. Secondary Outcome: Basal:Bolus Insulin Ratio
Description: Basal:Bolus Insulin Ratio.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Basal:Bolus Ratio
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 53
Basal:Bolus Ratio
  Baseline | 0.9 [0.7 to 1.2] | 0.8 [0.6 to 1.2] | 0.88 [0.69 to 1.27]
  At 13-week Follow Up | 1.0 [0.8 to 1.2] | 0.9 [0.6 to 1.3] | 0.96 [0.71 to 1.32]

36. Secondary Outcome: Weight
Description: Weight (kg)
Time Frame: 13 weeks
Population: Data not available in all participants.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
kg
  Baseline | 77.2 [66.3 to 93.4] | 73.0 [65.5 to 87.8] | 74 [62 to 86]
  At 13-week Follow Up: number analyzed (Participants) | 54 | 55 | 54
  At 13-week Follow Up | 79.2 [65.9 to 93.4] | 72.8 [65.8 to 87.8] | 75 [64 to 87]

37. Secondary Outcome: BMI
Description: Body Mass Index (BMI) kg/m2
Time Frame: 13 weeks
Population: Data not available in all participants
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
kg/m^2
  Baseline | 25.7 [23.4 to 30.0] | 25.1 [22.6 to 28.5] | 26 [22 to 29]
  At 13-week Follow Up: number analyzed (Participants) | 54 | 55 | 54
  At 13-week Follow Up | 25.6 [23.3 to 29.2] | 25.1 [23.1 to 28.1] | 26 [23 to 28]

38. Other Pre Specified Outcome: Ketone Events Defined as Day With Ketone Level >1.0 mmol/L
Description: Ketone events defined as day with ketone level > 1.0 mmol/L
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 5 | 1 | 7

39. Other Pre Specified Outcome: CGM-measured Hypoglycemic Events (>15 Minutes With Glucose Concentration <54 mg/dL)
Description: CGM-measured hypoglycemic events (>15 minutes with glucose concentration <54 mg/dL).
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: event rate per week
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
event rate per week | 0.4 [0.1 to 0.9] | 0.5 [0.1 to 0.9] | 0.4 [0.2 to 0.8]

40. Other Pre Specified Outcome: CGM-measured Hyperglycemic Events (>15 Minutes With Glucose Concentration >300 mg/dL)
Description: CGM-measured hyperglycemic events (>15 minutes with glucose concentration >300 mg/dL).
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Event Rate per Week
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Event Rate per Week | 1.6 [0.5 to 3.1] | 2.3 [0.9 to 5.3] | 1.0 [0.6 to 3.3]

41. Other Pre Specified Outcome: Worsening of HbA1c From Randomization to 13 Weeks by >0.5%
Description: Worsening of HbA1c from randomization to 13 weeks by >0.5%.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Participants | 8 | 20 | 3

42. Other Pre Specified Outcome: Serious Adverse Events With a Possible or Greater Relationship to a Study Device (Including Anticipated and Unanticipated Adverse Device Effects)
Description: Serious adverse events with a possible or greater relationship to a study device (including anticipated and unanticipated adverse device effects).
Time Frame: 13 weeks
Measure: Number; unit: Events
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events | 0 | 0 | 0

43. Other Pre Specified Outcome: Adverse Device Effects (ADE) That do Not Meet Criteria for SAE
Description: Adverse device effects (ADE) that do not meet criteria for SAE.
Time Frame: 13 weeks
Measure: Number; unit: Events
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events | 0 | 0 | 0

44. Other Pre Specified Outcome: Other Serious Adverse Events Not Related to a Study Device
Description: Other serious adverse events not related to a study device.
Time Frame: 13 weeks
Measure: Number; unit: Events
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events | 0 | 0 | 0

45. Other Pre Specified Outcome: Severe Hypoglycemic Events
Description: Number of Severe Hypoglycemic events over initial 13 weeks of trial
Time Frame: 13 weeks
Measure: Number; unit: Events
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events | 0 | 0 | 0

46. Other Pre Specified Outcome: Severe Hypoglycemic Event Rate Per 100 Person-years
Description: Number of severe hypoglycemic events per 100 person-years over initial 13 weeks of trial
Time Frame: 13 weeks
Measure: Number; unit: Events per 100 person-years
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events per 100 person-years | 0 | 0 | 0

47. Other Pre Specified Outcome: Diabetic Ketoacidosis (DKA) Events
Description: Number of DKA events over initial 13 weeks of trial
Time Frame: 13 weeks
Measure: Number; unit: Events
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events | 0 | 0 | 0

48. Other Pre Specified Outcome: Diabetic Ketoacidosis (DKA) Event Rate Per 100 Person-years
Description: Number of DKA events per 100 person-years over initial 13 weeks
Time Frame: 13 weeks
Measure: Number; unit: Events per 100 person-years
Groups:
- Closed Loop Control (CLC): PParticipants randomized to the closed loop control (CLC) arm will use the t:slim X2 with Control-IQ Technology & Dexcom G6 CGM for 3 months. Participants in this arm had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm are analyzed as part of the Objective 1 of the trial to compare CLC vs PLGS for 3 months following the use of 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial).
  Participants in this arm will continue to use CLC through commercial availability of the device after completion of the 3 months extension (Objective 3 of the trial).
- Predictive-Low Glucose Suspend (PLGS): PParticipants randomized to Predictive-Low Glucose Suspend (PLGS) arm will use the t:slim X2 with Basal-IQ & Dexcom G6 CGM for 3 months. Participants in this arm had 6 months of CLC in the primary trial (DCLP3 Pivotal Trial). Participants in this arm are analyzed as part of the Objective 1 of the trial to compare CLC vs PLGS for 3 months following the use of 6 mos of CLC in the primary trial (DCLP3 Pivotal Trial).
  Participants in this arm will use CLC through commercial availability of the device after the 3 months extension (Objective 3 of the trial).
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events per 100 person-years | 0 | 0 | 0

49. Other Pre Specified Outcome: Any Adverse Event Rate Per 100 Person-years
Description: Number of adverse events per 100 person-years over initial 13 weeks
Time Frame: 13 weeks
Measure: Number; unit: Events per 100 person-years
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
Number analyzed (Participants) | 54 | 55 | 55
Events per 100 person-years | 0 | 22.2 | 14.6

50. Other Pre Specified Outcome: Time in Target Range From Months 4-12
Description: CGM time in target range 70-180mg/dL for all participants using CLC from Months 4-12.
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage time in range
Groups:
- Closed-Loop Control (CLC) From 3 Months Until Study End: After 3 months, all participants continued or transitioned to Closed-Loop Control until study end. Specifically the initial 3 groups transitioned into one group using CLC: 1) CLC group continued CLC; 2) PLGS group transitioned to CLC and 3) the SAP to CLC group continued CLC. The timing of study end was not a fixed duration per participant and occurred following commercialization of device.
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage time in range | 68.8 (12.4)

51. Other Pre Specified Outcome: CGM Time Above 180 From Months 4-12
Description: CGM-measured % above 180mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 30 (13)

52. Other Pre Specified Outcome: CGM Mean Glucose From Months 4-12
Description: CGM-measured mean glucose from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
mg/dL | 161 (21)

53. Other Pre Specified Outcome: CGM Time Below 70 From Months 4-12
Description: CGM-measured % below 70 mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 1.38 (0.98)

54. Other Pre Specified Outcome: CGM Time Below 54 From Months 4-12
Description: CGM-measured % time below 54mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 0.17 [0.08 to 0.35]

55. Other Pre Specified Outcome: CGM Time in Range 70-140 mg/dL From Months 4-12
Description: CGM-measured % time in range 70-140mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 43.6 (11.4)

56. Other Pre Specified Outcome: Coefficient of Variation From Months 4-12
Description: CGM measured glucose variability measured with the coefficient of variation from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage SD of mean
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage SD of mean | 34 (5)

57. Other Pre Specified Outcome: Standard Deviation From Months 4-12
Description: CGM measured glucose variability measured with the standard deviation (SD) from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
mg/dL | 56 (14)

58. Other Pre Specified Outcome: CGM Time Below 60 From Months 4-12
Description: CGM-measured % below 60mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 0.37 [0.17 to 0.7]

59. Other Pre Specified Outcome: LBGI From Months 4-12
Description: LBGI from Months 4-12. Low blood glucose index by CGM with higher index indicating higher risk of hypoglycemia. Values <1 suggest minimal risk. Index of risk of low blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Gonder-Frederick LA, Young-Hyman D, Schlundt D, Clarke WL: Assessment of risk for severe hypoglycemia among adults with IDDM: validation of the low blood glucose index. Diabetes Care 21:1870-1875, 1998)
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
index | 0.45 (0.25)

60. Other Pre Specified Outcome: HBGI From Months 4-12
Description: HBGI from Months 4-12. High blood glucose index by CGM with higher values indicating higher risk of hyperglycemia. Index of risk of high blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Kumar A, Gonder-Frederick L, Clarke WL. Algorithmic evaluation of metabolic control and risk of severe hypoglycemia in type 1 and type 2 diabetes using self-monitoring blood glucose data. Diabetes Technol Ther 2003;5:817-828pmid:14633347)
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
index | 7.1 (3.8)

61. Other Pre Specified Outcome: CGM Hypoglycemia Events From Months 4-12
Description: CGM-measured events of at least 15 consecutive minutes <70mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: Events per Week
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
Events per Week | 2.9 (1.9)

62. Other Pre Specified Outcome: CGM Time >250 From Months 4-12
Description: CGM-measured % time >250 mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 8.9 (8.4)

63. Other Pre Specified Outcome: CGM Time >300 From Months 4-12
Description: CGM-measured % time >300 mg/dL from Months 4-12
Time Frame: Months 4-12
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
percentage of time | 3.5 (5.0)

64. Other Pre Specified Outcome: HbA1c at Month 6
Description: HbA1c measured at Month 6 of this extension study
Time Frame: Month 6 of study
Measure: Mean (Standard Deviation); unit: % of glycated hemoglobin
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 160
% of glycated hemoglobin | 7.04 (0.76)

65. Other Pre Specified Outcome: HbA1c at Month 9
Description: HbA1c measured at month 9 of this extension study
Time Frame: Month 9 of study
Measure: Mean (Standard Deviation); unit: % of glycated hemoglobin
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 157
% of glycated hemoglobin | 6.95 (0.8)

66. Other Pre Specified Outcome: HbA1c at Month 12
Description: HbA1c measured at Month 12 of this extension study
Time Frame: Month 12 of study
Measure: Mean (Standard Deviation); unit: % of glycated hemoglobin
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 102
% of glycated hemoglobin | 6.92 (0.74)

67. Other Pre Specified Outcome: Ketone Events Defined as Days With Ketone Level >1.0 mmol/L From Months 4-12
Description: Ketone Events Defined as Number of Days with at least one Ketone Level >1.0 mmol/L from Months 4-12
Time Frame: Months 4-12
Measure: Number; unit: days
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
days | 38

68. Other Pre Specified Outcome: CGM-measured Hypoglycemia Events (>15 Minutes With Glucose Concentration <54mg/dL) From Months 4-12
Description: CGM-measured Hypoglycemia Events (>15 minutes with glucose concentration <54mg/dL) from Months 4-12 measured as a rate per week.
Time Frame: Months 4-12
Measure: Median (Inter-Quartile Range); unit: Events per Week
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
Events per Week | 0.3 [0.1 to 0.7]

69. Other Pre Specified Outcome: CGM-measured Hyperglycemic Events From Months 4-12
Description: CGM-measured Hyperglycemic Events (>15 consecutive minutes with CGM glucose >300mg/dL) from Months 4-12
Time Frame: Months 4-12
Measure: Median (Inter-Quartile Range); unit: Event rate per week
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
Event rate per week | 1.5 [0.8 to 4.0]

70. Other Pre Specified Outcome: Number of Severe Hypoglycemic Events From Months 4-12
Description: Number of Severe Hypoglycemic Events from Months 4-12.
Time Frame: Months 4-12
Measure: Number; unit: events
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
events | 4

71. Other Pre Specified Outcome: Number of Diabetic Ketoacidosis (DKA) Events From Months 4-12
Description: Number of Diabetic Ketoacidosis (DKA) events from Months 4-12.
Time Frame: Months 4-12
Measure: Number; unit: events
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
events | 3

72. Other Pre Specified Outcome: Other Serious Adverse Events Not Related to a Study Device From Months 4-12
Description: Other Serious Adverse Events Not Related to a Study Device from Months 4-12.
Time Frame: Months 4-12
Measure: Number; unit: events
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
events | 4

73. Other Pre Specified Outcome: Any Adverse Event Rate Per 100 Person-years From Months 4-12
Description: Any Adverse Event Rate per 100 person-years from Months 4-12.
Time Frame: Months 4-12
Measure: Number; unit: events rate per 100 person-years
Arm/Group | Closed-Loop Control (CLC) From 3 Months Until Study End
Number analyzed (Participants) | 161
events rate per 100 person-years | 39

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Closed Loop Control (CLC) | Predictive-Low Glucose Suspend (PLGS) | SAP to CLC Group
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/54 | 3/55 | 2/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Loop Control (CLC) (N=54) | Predictive-Low Glucose Suspend (PLGS) (N=55) | SAP to CLC Group (N=55)
Hyperglycemia or ketosis events without meeting criteria for Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03591354/Prot_002.pdf
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT03591354/SAP_001.pdf